CLINICAL TRIAL: NCT00624533
Title: Evaluation of the Efficiency of Physiotherapeutic Treatment of Non-Specific Low Back Pain in Primary Care Centers Through GDS Techniques for Articular and Muscular Chains
Brief Title: Efficiency of GDS Method for Lumbar Stabilization for Non-Specific Low Back Pain in Primary Care
Acronym: GDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carlos III Health Institute (Other Government)
Collaborators: Agencia Lain Entralgo (Other Government); Public Health Service of Madrid (Other)
Responsible Party: Joaquín Arenas Barbero, Carlos III Health Institute. General Director for evaluation and research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI051650; PI051650; LA2007PISINISCIII77
Record Dates: First submitted 2008-02-19; First posted 2008-02-27 (Estimated); Last update posted 2008-02-27 (Estimated); Status verified 2008-02

CONDITIONS: Low Back Pain
Keywords: Low back Pain; Physical Therapy Modalities; Exercise Movement Techniques; Primary Health Care
MeSH Terms: conditions — Low Back Pain | interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Primary Health Care Conventional Physiotherapy Treatment (based in electrotherapy)
  Interventions: Behavioral: Conventional Physical Therapy in Primary Health Care
- B (Experimental): Group B was treated with the GDS Method (muscular and articular chains physiotherapy method)
  Interventions: Behavioral: GDS Method (muscular chains physical therapy method)

INTERVENTIONS:
Behavioral: GDS Method (muscular chains physical therapy method) — Experimental group received 15 GDS method sessions based on the equilibration of articular and muscular tensions that reduced trunk and lumbopelvic stability. GDS method combine specific technics of manual therapy, spinal stabilisation and stretching exercises (4 sessions),supervised group exercise therapy (10 sessions) and home exercise programme with individualised exercises (1 session) Experimental group received 2 sessions of 50 minutes per week during 8 weeks.
  Arms: B
Behavioral: Conventional Physical Therapy in Primary Health Care — Conventional Physical Therapy in Spanish Primary Care Units are based on Electrotherapy (TENS and microwave thermotherapy) and a standard written advices. Patients received 14 sessions of 40 minutes of conventional TENS, 10 minutes of microwave thermotherapy and 1 last session of standard written advices.
  Conventional Physical Therapy group received 2 sessions of 50 minutes per week during 8 weeks.
  Arms: A

SUMMARY:
The purpose of this randomized controlled trial was to assess the effectiveness of GDS Treatment Method for patients with subacute or chronic non-specific low back pain in Primary Care of Spanish National Health Service.

DETAILED DESCRIPTION:
Low back pain is one of the most frequent ailments in industrialized countries, with a lifetime prevalence of more than 70%. It is responsible for a major portion of work absenteeism and is actually among those conditions which generate the greatest expense due to health and labor costs.

The Spanish National Health Service is a universal and free health care system. Non-specific low back pain (LBP) is a prevalent disorder, generating large health and social costs.

There is considerable variation in LBP related clinical practice and a considerable number of clinical guidelines have been developed for the management of subacute and chronic LBP patients.

Experience in Primary Care Centers of Madrid shows that physiotherapeutic intervention based on GDS Method for Articular and Muscular Chains is an efficient technique in the treatment of patients with diagnosis of non-specific low back pain compared with conventional physiotherapy treatment in Primary Care based on electrotherapy (TENS and microwave)

Currently, no randomized studies examining the effects of this method for patients with subacute or chronic non-specific low back pain have been published.

ELIGIBILITY:
Inclusion Criteria:

Participants were required to:

* Be aged 18 years or older;
* Have been diagnosed with simple mechanical LBP by their doctor and prescribed physiotherapy;
* Have an impairment secondary to functional overload and/or poor postural habits (patients with certain occupations were excluded if these could act as confounding factors);
* Not be receiving any other form of treatment;
* Not be neurologically compromised; and
* To be in a subacute or chronic stage of LBP exceeding 4 weeks.

Exclusion Criteria:

Subjects were excluded if they:

* Showed clear symptoms of depression;
* Refused to participate;
* Did not sign the informed consent form;
* Had any cognitive impairment that would prevent them from following instructions;
* Were unable to understand Spanish sufficiently to adequately follow instructions;
* Had the intention of moving from the area;
* Had any form of contraindication to the physiotherapeutic techniques to be applied to both groups;
* Had red flags, or warning signs, of serious illness such as cancer, infection, fracture or cauda equinal syndrome;
* Had yellow flags, or risk factors, for a psychological disorder or had lumbar pain whose main cause was not mechanical.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-01; Primary Completion 2006-03 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Intensity of pain (VAS) | At baseline, immediately after intervention,at 3-months and 6-months

SECONDARY OUTCOMES:
Disability (Oswestry questionnaire) Quality of life (SF-36 questionnaire) Elasticity goniometric test for lumbopelvic region | At baseline, immediately after intervention,at 3-months and 6-months

CONTACTS AND LOCATIONS:
Overall Officials: José L Chicharro, MD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Complutense University, Madrid, Spain/Madrid, Spain

REFERENCES:
- [Background] Kovacs FM, Abraira V, Zamora J, Teresa Gil del Real M, Llobera J, Fernandez C, Bauza JR, Bauza K, Coll J, Cuadri M, Duro E, Gili J, Gestoso M, Gomez M, Gonzalez J, Ibanez P, Jover A, Lazaro P, Llinas M, Mateu C, Mufraggi N, Muriel A, Nicolau C, Olivera MA, Pascual P, Perello L, Pozo F, Revuelta T, Reyes V, Ribot S, Ripoll J, Ripoll J, Rodriguez E; Kovacs-Atencion Primaria Group. Correlation between pain, disability, and quality of life in patients with common low back pain. Spine (Phila Pa 1976). 2004 Jan 15;29(2):206-10. doi: 10.1097/01.BRS.0000107235.47465.08. PMID 14722416